CLINICAL TRIAL: NCT06054230
Title: Genomic Sequencing for Evaluation of Fetal Structural Anomalies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-36483
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fetal Structural Anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Genomic Sequencing (Experimental)
  Interventions: Device: Genomic Sequencer

INTERVENTIONS:
Device: Genomic Sequencer — Genomic Sequencing Device

SUMMARY:
This study follows an observational prospective cohort design. Women with fetal structural anomalies are routinely offered diagnostic testing with chorionic villus sampling or amniocentesis, with analysis for chromosomal analysis using karyotype or microarray analysis. Women in whom such testing does not explain the fetal phenotype, or in whom a genetic disease is strongly suggested based on the phenotype or a pattern of recurrent anomalies, will be offered exome sequencing (ES) and/or genome sequencing (GS) through the UCSF CLIA certified Genomic Medicine Laboratory. In advance of study enrollment, patients have been counseled regarding the structural anomalies in the fetus and offered pregnancy termination. The sequencing results for on-going pregnancies have a turnaround time of 2-4 weeks, and in the majority of cases are available after decisions have been made regarding continuation or termination of pregnancy.

Patients who decline diagnostic testing but who have a prenatally identified anomaly may be offered the option of testing on umbilical cord blood at delivery or on the placenta or other products of conception after a stillbirth or pregnancy termination. The project is exploratory in nature, with the ultimate goal of contributing to a growing body of phenotypic data and understanding how providers and patients utilize genomic (either exome or genome) sequencing results during pregnancy.

DETAILED DESCRIPTION:
Over the last several years, UCSF providers in the Fetal Treatment Center (FTC) and Prenatal Diagnosis Center (PDC) have been conducting genomic sequencing research studies for prenatal cases of fetal structural anomalies and pregnancy complications. This study seeks to build on preliminary work by our team at UCSF.

The investigators will study:

A. The effectiveness of sequencing as a tool for diagnosing the underlying genetic cause in fetuses with structural anomalies B. The prenatal presentation of genetic diseases and how genetic variants may be associated with specific fetal phenotypes C. How identifying a genetic diagnosis can help providers predict prognosis, counsel patients, and provide focused antenatal and postnatal management of the fetus/infant D. How patients and families understand and benefit from identifying an underlying genetic diagnosis in a pregnancy with fetal structural anomalies

Specific Aims:

A. Demonstrate the effectiveness of sequencing as a tool for diagnosing the underlying genetic cause in fetuses with structural anomalies B. Define the prenatal presentation of genetic diseases and how genetic variants may be associated with specific fetal phenotypes C. Determine how identifying a genetic diagnosis can help providers predict prognosis, counsel patients, and provide focused antenatal and postnatal management of the fetus/infant D. Identify how patients and families understand and benefit from identifying an underlying genetic diagnosis in a pregnancy with fetal structural anomalies

This study follows an observational prospective cohort design. Patients with fetal structural anomalies are routinely offered diagnostic testing with chorionic villus sampling or amniocentesis. Patients in whom such testing does not explain the fetal phenotype, or in whom a genetic disease is strongly suggested based on the phenotype or a pattern of recurrent anomalies, will be offered exome sequencing (ES) and/or genome sequencing. Patients who decline prenatal diagnostic testing but who have a prenatally identified anomaly may be offered the option of testing on umbilical cord blood at delivery or on the placenta or other products of conception after a stillbirth or pregnancy termination. Blood or saliva samples will be collected on both parents, when possible, to allow the option of trio ES/GS or for follow up Sanger sequencing on these specimen determining inheritance of any potentially significant fetal variants that are identified. Patients will be asked to accept or decline analysis for secondary findings, as recommended by the American College of Medical Genetics and Genomics.Exome and genome sequencing will be performed in the UCSF clinical Genomic Medicine Laboratory, and patients will receive results through the CLIA certified clinical laboratory. Patients will be managed as per usual clinical protocols. Clinical data will be collected regarding the pregnancy, delivery, neonatal and early childhood outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant individual >18 years of age
2. Pregnant with a fetus (singleton or multiple gestation) affected by one or more fetal anomalies, unexplained fetal death after 14 wks, unexplained severe fetal growth restriction (< 3%ile), unexplained severe polyhydramnios

Exclusion Criteria:

1. Declines diagnostic testing with karyotype or microarray
2. Fetal anomaly explained by other testing (viral infection, aneuploidy or copy number variant detected by microarray)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2030-07-15 (Estimated); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of prenatal genomic sequencing | Up to three months
  Number of cases with a positive finding among all cases tested

CONTACTS AND LOCATIONS:
Overall Officials: Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No